CLINICAL TRIAL: NCT05301816
Title: A Post-Market, Multicenter, Prospective, Global Clinical Study to Evaluate the Real-world Experience of Spinal Cord Stimulation That Includes 10 kHz in the Management of Chronic Intractable Pain Associated With Diabetic Neuropathy.
Brief Title: PDN Post Market, Multicenter, Prospective, Global Clinical Study
Acronym: PDN-PM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nevro Corp (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA2021-03 INT PDN-PM
Record Dates: First submitted 2022-02-11; First posted 2022-03-31 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Neuropathy, Painful
Keywords: Spinal Cord Stimulation (SCS)
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- IPG Activated (Experimental): The group of participants who have had a successful trial (>50% pain relief) during the trial phase
  Interventions: Device: Spinal Cord Stimulator (SCS)

INTERVENTIONS:
Device: Spinal Cord Stimulator (SCS) — Spinal cord stimulation system (SCS) is an approved system to manage chronic intractable pain of the limbs and/or leg by delivering electrical stimulation using implantable leads and rechargeable implantable pulse generator (IPG) with 16 output channels. The IPG is implanted in a subcutaneous pocket and is capable of stimulating the spinal cord nerves when used with one or two 8-contact percutaneous or paddle leads.

SUMMARY:
The purpose of this post-market study is to evaluate the real-world experience of Nevro's Spinal Cord Stimulation (SCS) therapy in patients with chronic, intractable leg pain due to painful diabetic neuropathy (PDN). This is a multicenter, prospective, observational global study, that will partner diabetes management teams with pain physicians to provide an interdisciplinary treatment regimen for PDN patients. Outcomes will be assessed via standardized assessments.

ELIGIBILITY:
Inclusion Criteria:

To participate in the study, patients must meet all the following inclusion criteria:

1. Have been clinically diagnosed with diabetes, according to the local country diabetes association guidelines, as well as painful diabetic neuropathy (PDN) of the lower limbs refractory to conventional medical management.
2. Average pain intensity (over the last 7 days) of ≥5 out of 10 cm on the Visual Analog Scale (VAS) in the lower limbs at enrollment/baseline.
3. The clinical decision has been made to provide treatment using the Nevro Spinal Cord Stimulation that includes 10 kHz therapy prior to enrollment in the study.
4. Be willing and capable of giving written informed consent.
5. Be willing and able to comply with study-related requirements and procedures and attend all scheduled visits.

Exclusion Criteria:

To participate in the study, patients must not meet any of the following exclusion criteria:

1. Have a diagnosis of a lower limb mononeuropathy (e.g., causalgia and tibial or peroneal neuropathies), have had a lower limb amputation other than toes, or have large (≥3 cm) and/or gangrenous ulcers of the lower limbs
2. Have a medical condition or diagnosis that is inconsistent with Nevro's SCS System guidelines in the Physician's Manual for the relevant country, or as per standard clinical practice.
3. Have a medical condition or pain in other areas, not intended to be treated in this study, that could interfere with study procedures, accurate pain reporting, and/or confound the evaluation of study endpoints, as determined by the Investigator (such as primary headache, fibromyalgia, post-herpetic neuralgia, osteoarthritis, peripheral vascular disease, or small vessel disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 497 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Trial success rate/Responder rate | 2 weeks
  Percentage of patients with a successful trial phase (responder rate) i.e. at least 50% reduction in patient-reported overall pain relief.
Patient-reported overall pain relief | 12 months
  The average percentage of patient-reported pain relief at 3,6 and 12 months.
Leg pain | 12 months
  Leg pain will be assessed using a 10 cm Visual Analog Scale (VAS) with 0 indicating no pain and 10 indicating the worst pain. Following outcome measures will be derived from the VAS score on leg pain.
  * Responder rate for leg pain i.e. percentage of patients who experience at least 50% reduction in leg pain compared to Baseline at 3, 6, and 12 months.
  * Change from Baseline in mean leg pain at 3, 6, and 12 months
  * Percentage change from Baseline in mean leg pain at 3, 6, and 12 months
Quality of life measure | 12 months
  Change from baseline in quality of life at 3, 6 and 12 months will be assessed using the EQ-5D-5L questionnaire.
Pain Inventory | 12 months
  Change from baseline in pain symptoms at 3, 6 and 12 months assessed by 11-point BPI-DPN (Brief Pain Inventory for Diabetic Peripheral Neuropathy) pain scale, with 0 indicating no pain and 10 indicating worst pain.
Global impression of change in health status | 12 months
  The patient's general health status at 3, 6 and 12 months will be assessed both by the patients themselves as well as the study investigators using the 7-point PGIC (Patient Global Impression of Change) and the CGIC (Clinician Global Impression of Change) instrument respectively. Responses for this questionnaire range from "no change (or condition has got worse)" to "a great deal better".

OTHER OUTCOMES:
Patients Work Status | 12 months
  Patients' current work status (working for pay, working without pay, self-employed, out of work for more than 1 year, out of work for less than 1 year, homemaker/taking care of the house and/or family, student, retired, unable to work) will be collected at baseline and repeated at the 12 months follow up visit.
Device Safety | 12 months
  Subjects will be assessed for the procedure and device-related adverse events starting at enrollment and continuing through study completion. An adverse event may include but is not limited to infection, lead revisions, IPG revisions, device malfunction, and explantation of devices.

CONTACTS AND LOCATIONS:
Overall Officials: David Caraway, MD, Study Director — Chief Medical Officer, Nevro Corp
Locations (8):
- United States (8):
  - Neuroversion, Inc., Anchorage, Alaska
  - Michigan Pain Specialists, Ann Arbor, Michigan
  - Henry Ford Health, West Bloomfield, Michigan
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Clinical Investigations, LLC, Edmond, Oklahoma
  - Columbia Pain Management, Milwaukie, Oregon
  - WellSpan Interventional Pain Specialists, York, Pennsylvania
  - Virginia Interventional Pain & Spine Centers, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No